CLINICAL TRIAL: NCT04582929
Title: 24-Week Prospective, Double-Blinded, Randomized, Cross-over Design in Multicenter Study of 50 Unit of Neubotulinum Toxin Type A (Neuronox) and 100 Unit of Neubotulinum Toxin Type A (Neuronox) Injection for Cervical Dystonia in Thai Patients
Brief Title: Neubotulinum Toxin Injection in Cerivical Dystonia
Acronym: NTCD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Principal Investigator, Dr Subsai Kongsaengdao, Associate Professor Subsai Kongsaengdao, Department of Medical Services Ministry of Public Health of Thailand
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-02-2020
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Double Blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: complete Double Blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 unit of Neubotulinum Toxin Type A (Neuronox) (Experimental): 50 unit of Neubotulinum Toxin Type A (Neuronox) injection for Cervical Dystonia in patient diagnosed with cervical dystonia according to clinical diagnosis
  Interventions: Drug: Neuronox ® Injection
- 100 unit of Neubotulinum Toxin Type A (Neuronox) (Experimental): 100 unit of Neubotulinum Toxin Type A (Neuronox) injection for Cervical Dystonia in patient diagnosed with cervical dystonia according to clinical diagnosis
  Interventions: Drug: Neuronox ® Injection

INTERVENTIONS:
Drug: Neuronox ® Injection — Neuronox ® 50 or 100 unit intramuscular injection
  Other Names: Neuronox ® 50 unit or 100 unit

SUMMARY:
24-Week Prospective, Double-Blinded, Randomized, Cross-over design in Multicenter Study of 50 unit of Neubotulinum Toxin Type A (Neuronox) and 100 unit of Neubotulinum Toxin Type A (Neuronox) injection for Cervical Dystonia in patient diagnosed with cervical dystonia according to clinical diagnosis. It was designed to evaluate the efficacy, safety, tolerability, quality of life and the comparesion the improvement after treatment by of 50 unit of Neubotulinum Toxin Type A (Neuronox) and 100 unit of Neubotulinum Toxin Type A (Neuronox) injection.

DETAILED DESCRIPTION:
Three documented studies showed the clinical use of botulinum toxin for migraine prophylaxis.(26) Neubotulinum Toxin Type A, (Neu-BoNT/A), (Neuronox® ) (Medytox Inc, Ochang-eup, Cheongwon-gu, Cheongju-si, Chungcheongbuk-do, Republic of Korea), also known as Meditoxin in Korea, is a newly manufactured BoNT-A (Neu-BoNT/A) that was developed to provide features close to onabotulinum toxin A (5). Neuronox was tested in a murine model, and its effect on muscle force generation was equivalent to Botox® (ona-BoNT/A) (6). A previous multicenter randomized controlled trial showed that Neuronox and Botox® have equivalent efficacy and safety for the treatment of spastic equinus in children with cerebral palsy (6). However, 50 unit of Neubotulinum Toxin Type A (Neuronox) and 100 unit of Neubotulinum Toxin Type A (Neuronox) has not yet been investigated in cervical dystonia. This study is the extension of the NCT03805152

ELIGIBILITY:
Inclusion Criteria:

•The subject has to grant permission to enter into the study by signing and dating the informed consent form before completing any study-related procedure such as any assessment or evaluation not related to the normal medical care of the subject.

Able to give written inform consent and retained one copy of the consent form

* Male or female subject, aged between 18 - 100 years old.
* Subject diagnosed to be cervical dystonia.
* Female subject in good health and sexually active was instructed by the investigator to avoid pregnancy during the study and to use condom or other contraceptive measure if necessary. The subject was required to have a negative urine pregnancy test before being eligible for the study. (At each of the subsequent visit, a urine pregnancy test was performed).
* Subject judged to be reliable for compliance for taking medication and capable of recording the effects of the medication and motivated in receiving benefits from the treatment.
* Subject should undergo a normal physical and neurological examination TWSTRS, CDIP-58, SF36, and CES-D • during the whole study period

Exclusion Criteria:

* The subject was pregnant or lactating.
* The subject was a female at risk of pregnancy during the study and not taking adequate precautions against pregnancy.
* The subject had a known hypersensitivity to any of the test materials or related compounds.
* The subject was unable or unwilling to comply fully with the protocol.
* The subject received any unlicensed drug within the previous 6 months.
* Treatment with investigational drug (s) within 6 months before the screening visit. • The subject had previously entered in this study.

Subject with past history of botulism, other neuromuscular disorder (e.g. myasthenia gravis, Lambert - Elton Syndrome)

* Subject with significant medical / neurological / psychiatric disorders such as blood dyscrasia, thrombocytopenia, rheumatoid arthritis, congestive heart failure, coronary artery heart diseases, dementia, psychosis, or other conditions which could influence the clinical trial.
* Known history of drug abuse (narcotic (s), cafergot, or others) or drug (botulinum toxin type A) allergy.
* Unable to cooperate fill-up TWSTRS, CDIP-58, SF36, and CES-D • Patient who planned to schedule elective surgery during the study.
* The used of aminoglycoside antibiotics and curare were not allowed during the study.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating scale ( TWSTRS) | 24 week
  WSTRS ranged( 0-85 by summation of all 3 sub- scales ) higher represent a worse outcome TWSTRS Sub- scale includes
  TWSTRS-Total severity scale ( maximum 35 points) TWSTS-Disability scale (maximum 30 points) TWSTS-Pain scale (maximum 20 points)
Cervical Dystonia Impact Profile 58 ( CDIP-58) | 24 week
  Cervical Dystonia Impact Profile-58 items composed of 8 sub-scale Total score by summation of 8 subscale higher represent a worse outcome Analysis both total score (range 58-290 points) And sub-scale analysis composed of Head and neck symptoms ( 6 items ; 6-30 points) Pain and discomfort ( 5 items ; 5-25 points) Upper limb activity ( 9 items ; 9-45 points) Walking ( 9 items ; 9-45 points) Sleep ( 4 items ; 4-20 points) Annoyance ( 8 items ; 8-40 points) Mood (7 items ; 7-35 points) Psychosocial functioning ( 10 items ; 10-50 points)

SECONDARY OUTCOMES:
Comparesion the quality of life 36 item ( SF 36) | 24 week
  Comparesion the quality of life (SF 36) pre- and post- 12 and 24 week ttreatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) this score has special formula calculation
Depression scale measured by Center of Epidemiologic Study of Depression 20 item ( CES-D 20) | 24 week
  Comparesion of CES-D pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) Score ranged from 20-80 points higher represent a worse outcome
Depression scale measured by Patient Health Questionnaire Depression Scale (PHQ-9) | 24 week
  Comparesion of PHQ-9 pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) There is the special scale calculation for diagnosis Major depressive disorder, Other depressive disorder and others,higher points /score represent a worse outcome ranged 0-27 points plus 3 points Total summation of 5-9 points indicate Minimal symptoms, 10-14 Minor depression ++ or Dysthymia* or Major depression, mild , 15-19 points Major depression, moderately severe
  ≥ 20 Major depression, severe (range PHQ 9 0-27 ) higher represent a worse outcome
Clinical Global Impression of Changed ( CGIC) | 24 week
  Comparesion of CGIC pre- and post- 12 and 24 week treatment with 50 unit of Neubotulinum Toxin Type A (Neuronox) and 250 unit of Abobotulinum Toxin Type A (Dysport) (range -3 to 3 points: -3,-2,-1,0,1,2,3)

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Rajavithi Hospital, Bangkok
  - Lampang Hospital, Lampang
  - Suratthani Hospital, Surat Thani
  - Sappasitthiprasong Hospital, Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kongsaengdao S, Maneeton B, Maneeton N. Quality of life in cervical dystonia after treatment with botulinum toxin A: a 24-week prospective study. Neuropsychiatr Dis Treat. 2017 Jan 10;13:127-132. doi: 10.2147/NDT.S116325. eCollection 2017. PMID 28138245
- [Result] Kongsaengdao S, Maneeton N, Maneeton B. Long-term quality of life in cervical dystonia after treatment with abobotulinum toxin A: a 2-year prospective study. Neuropsychiatr Dis Treat. 2018 Apr 26;14:1119-1124. doi: 10.2147/NDT.S152252. eCollection 2018. PMID 29731634